CLINICAL TRIAL: NCT02626715
Title: A Phase II Study of Myeloablative and Reduced-Intensity Conditioning Regimens for Children and Young Adults With Acute Myeloid Leukemia or Myelodysplastic Syndrome Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Reduced-Intensity Conditioning (RIC) and Myeloablative Conditioning (MAC) for HSCT in AML/MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Randy Windreich (Other)
Responsible Party: Sponsor-Investigator, Randy Windreich, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19030327
Record Dates: First submitted 2015-09-24; First posted 2015-12-10 (Estimated); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Hematopoietic Stem Cell Transplant (HSCT)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Alemtuzumab; Hydroxyurea; fludarabine phosphate; Melphalan; Thiotepa; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced-Intensity Conditioning (Active Comparator): Campath (alemtuzumab), Droxia (hydroxyurea), Fludara (fludarabine), Alkeran (melphalan), Thiotepa (triethylenethiophosphoramide)
  Trade Name (generic name)
  Interventions: Drug: Reduced-Intensity Conditioning Regimen
- Myeloablative Conditioning (Active Comparator): Campath (alemtuzumab), Thiotepa (triethylenethiophosphoramide) , Fludara (fludarabine), Busulfex (busulfan)
  Trade Name (generic name)
  Interventions: Drug: Myeloablative Conditioning Regimen

INTERVENTIONS:
Drug: Reduced-Intensity Conditioning Regimen — Campath (alemtuzumab) - drug class: monoclonal antibody Droxia (hydroxyurea) - drug class: antimetabolite Fludara (fludarabine) - drug class: antimetabolite Alkeran (melphalan) - drug class: alkylating agent Thiotepa (triethylenethiophosphoramide) - drug class: cytotoxic agent
  Other Names: Campath, Droxia, Fludara, Alkeran, Thiotepa
  Arms: Reduced-Intensity Conditioning
Drug: Myeloablative Conditioning Regimen — Campath (alemtuzumab) - drug class: monoclonal antibody Thiotepa (triethylenethiophosphoramide) - drug class: cytotoxic agent Fludara (fludarabine) - drug class: antimetabolite Busulfex (busulfan) - drug class: alkylating agent
  Other Names: Campath, Thiotepa, Fludara, Busulfex
  Arms: Myeloablative Conditioning

SUMMARY:
The purpose of this study is to compare safety and efficacy of reduced-intensity conditioning and myeloablative conditioning regimens prior to HSCT in high-risk AML/MDS pediatric and young adult patients. This study investigates the use of two novel conditioning therapies for hematopoietic stem cell transplant (HSCT). The primary focus of both the investigators' myeloablative and reduced-intensity conditioning regimens is to reduce overall toxicity so that pediatric and young adult patients with high-risk AML/MDS with significant pretransplant comorbidities who would have been ineligible to proceed to HSCT previously can now receive potentially life-saving treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

Individuals must meet all the following criteria to be eligible for this study.

* Subject, parent, or legal guardian, if applicable, must have given written informed consent. For patients ≤ 17 years of age who are developmentally able, assent or affirmation will be obtained.
* Age 0-26, inclusive, at time of consent.
* Diagnosis of myelodysplastic syndrome or acute myeloid leukemia, either high-risk (defined below), relapsed or primary refractory, MRD-positive without circulating myeloblasts or active extramedullary disease at the time of transplant. Active marrow disease is permitted. High-risk AML features are defined by the following: RAM phenotype; adverse cytogenetic abnormalities of monosomy 5, monosomy 7, 5q deletion, or other unfavorable prognostic markers according to cytogenetics, FISH, or next generation sequencing (NGS); presence of FLT3 positive internal tandem duplication (FLT3/ITD+), particularly high allelic ratio; treatment-related AML; or positive minimal residual disease (MRD) at end of Induction I.
* Stem cell sources include bone marrow, peripheral blood stem cells, or umbilical cord blood. Related bone marrow, peripheral blood stem cell, or cord blood unit: sibling should be HLA-matched at A, B, and DR-B1 loci. Unrelated cord blood unit should be at a minimum of 4/6 matched at antigen level on HLA A and B, and allele level at HLA DR-B1 loci. Unrelated bone marrow or peripheral blood stem cell donor should be HLA allele level matched at DR-B1.
* Minimum pre-freezing cell dose for cord blood units: 3 x 10^7 total nucleated cells/kg and 1.5 x 10^5 CD34+ cells/kg. If this is not attainable, then double cord blood transplant should be considered.
* Subject must have adequate performance status: Lansky score ≥60% for patients <16 years, Karnofsky score ≥60% for patients ≥16 years.
* Subject must have adequate pre-transplant organ function to undergo one of the two conditioning regimens, either the myeloablative conditioning (MAC) OR reduced-intensity conditioning (RIC) regimen. If a subject does not meet the following organ function criteria for the MAC regimen, the RIC regimen will be considered if eligibility criteria is met. The RIC regimen may also be considered, regardless of MAC eligibility, if deemed appropriate by the Principal Investigator and/or treating physician.

Pre-transplant organ function criteria for Myeloablative Conditioning regimen:

* Renal: creatinine clearance or radioisotope GFR ≥70 mL/min/1.73 m2.
* Hepatic: total bilirubin ≤2.0 mg/dL unless the increase in bilirubin is attributable to Gilbert's syndrome; and SGOT (AST), SGPT (ALT), and Alkaline Phosphatase <4 x upper limit of normal (ULN) for age.
* Cardiac: normal cardiac function by echocardiogram or radionuclide scan, as defined by left ventricular ejection fraction at rest >45% or shortening fraction >26%.
* Pulmonary: FEV1, FVC, and DLCO (corrected for hemoglobin) ≥50% of predicted; if unable to perform pulmonary function tests, then oxygen saturation ≥92% on room air.

OR

Pre-transplant organ function criteria for Reduced-Intensity Conditioning regimen:

* Renal: creatinine clearance or radioisotope GFR ≥70 mL/min/1.73 m2.
* Hepatic: total bilirubin ≤2.5 mg/dL unless the increase in bilirubin is attributable to Gilbert's syndrome; and SGOT (AST), SGPT (ALT), and Alkaline Phosphatase <5 x upper limit of normal (ULN) for age.
* Cardiac: normal cardiac function by echocardiogram or radionuclide scan, as defined by left ventricular ejection fraction at rest >40% or shortening fraction >26%.
* Pulmonary: FEV1, FVC, and DLCO (corrected for hemoglobin) ≥40% of predicted; if unable to perform pulmonary function tests, then oxygen saturation ≥92% on room air.

  * HIV and HTLV negative, by either PCR or serology.
  * Negative pregnancy test for females ≥10 years old or who have reached menarche.
  * All females of childbearing potential and sexually active males must agree to use an FDA approved method of birth control for up to 12 months after HSCT or for as long as they are taking any medication that may harm a pregnancy, an unborn child or may cause a birth defect.

EXCLUSION CRITERIA:

Individuals who meet any of the following criteria are not eligible for this protocol.

* Uncontrolled bacterial, viral, fungal, or other infection at the time of cytoreduction, defined by positive blood cultures and/or fevers >38.0 within 24 hours of start of conditioning therapy.
* Females who are pregnant or who are lactating.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Additional Exclusion Criteria for Myeloablative Conditioning (MAC) Only Individuals who meet any of the following criteria are not eligible for the MAC regimen.

* Recipient of either an autologous or allogeneic stem cell transplant within 3 months of the start of conditioning.
* Patients with any inherited bone marrow failure syndrome including, but not limited to, Fanconi anemia, Shwachman-Diamond syndrome, dyskeratosis congenita or Down syndrome (defined as either constitutional trisomy 21 or constitutional mosaicism of trisomy 21).

Ages: 0 Months to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Windreich, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced-Intensity Conditioning: Conditioning Arm nonrandomly assigned based on eligibility (inclusion/exclusion) criteria.
  Campath (alemtuzumab), Droxia (hydroxyurea), Fludara (fludarabine), Alkeran (melphalan), Thiotepa (triethylenethiophosphoramide)
  Trade Name (generic name)
  Reduced-Intensity Conditioning Regimen: Campath (alemtuzumab) - drug class: monoclonal antibody Droxia (hydroxyurea) - drug class: antimetabolite Fludara (fludarabine) - drug class: antimetabolite Alkeran (melphalan) - drug class: alkylating agent Thiotepa (triethylenethiophosphoramide) - drug class: cytotoxic agent
- Myeloablative Conditioning: Conditioning Arm nonrandomly assigned based on eligibility (inclusion/exclusion) criteria.
  Campath (alemtuzumab), Thiotepa (triethylenethiophosphoramide) ,Fludara (fludarabine), Busulfex (busulfan)
  Trade Name (generic name)
  Myeloablative Conditioning Regimen: Campath (alemtuzumab) - drug class: monoclonal antibody Thiotepa (triethylenethiophosphoramide) - drug class: cytotoxic agent Fludara (fludarabine) - drug class: antimetabolite Busulfex (busulfan) - drug class: alkylating agent
Period: Overall Study
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Started | 6 | 15
Completed | 6 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Reduced-Intensity Conditioning: Campath (alemtuzumab), Droxia (hydroxyurea), Fludara (fludarabine), Alkeran (melphalan), Thiotepa (triethylenethiophosphoramide)
  Trade Name (generic name)
  Reduced-Intensity Conditioning Regimen: Campath (alemtuzumab) - drug class: monoclonal antibody Droxia (hydroxyurea) - drug class: antimetabolite Fludara (fludarabine) - drug class: antimetabolite Alkeran (melphalan) - drug class: alkylating agent Thiotepa (triethylenethiophosphoramide) - drug class: cytotoxic agent
- Myeloablative Conditioning: Campath (alemtuzumab), Thiotepa (triethylenethiophosphoramide) , Fludara (fludarabine), Busulfex (busulfan)
  Trade Name (generic name)
  Myeloablative Conditioning Regimen: Campath (alemtuzumab) - drug class: monoclonal antibody Thiotepa (triethylenethiophosphoramide) - drug class: cytotoxic agent Fludara (fludarabine) - drug class: antimetabolite Busulfex (busulfan) - drug class: alkylating agent
- Total: Total of all reporting groups
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning | Total
Number analyzed (Participants) | 6 | 15 | 21
Age, Continuous [Median (Full Range); unit: years] | 17.3 [9.7 to 18.9] | 8 [0.8 to 17.3] | 12.3 [0.8 to 18.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 13 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 13 | 18
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 14 | 20
  Puerto Rico | 0 | 1 | 1
Diagnosis [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia (AML) | 5 | 10 | 15
  Myelodysplastic syndrome (MDS) | 1 | 5 | 6
Stem Cell Source [Count of Participants; unit: Participants]
  Bone Marrow | 4 | 5 | 9
  Peripheral Blood | 0 | 3 | 3
  Umbilical Cord Blood | 2 | 7 | 9
Donor Source [Count of Participants; unit: Participants]
  Sibling donor | 4 | 2 | 6
  Unrelated donor | 2 | 13 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Non-relapsed Deaths by 100 Days Post-transplant in Pediatric Patients Receiving a Myeloablative or Reduced-intensity Preparative Regimen Prior to HSCT for High-risk AML and MDS.
Description: Number of non-relapsed deaths that occur
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Groups:
- Myeloablative Conditioning: Campath (alemtuzumab), Thiotepa (triethylenethiophosphoramide) ,Fludara (fludarabine), Busulfex (busulfan)
  Trade Name (generic name)
  Myeloablative Conditioning Regimen: Campath (alemtuzumab) - drug class: monoclonal antibody Thiotepa (triethylenethiophosphoramide) - drug class: cytotoxic agent Fludara (fludarabine) - drug class: antimetabolite Busulfex (busulfan) - drug class: alkylating agent
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 15
Participants | 1 | 0

2. Primary Outcome: Preliminary Efficacy (Event-free Survival at 6 Months) in Pediatric Patients Receiving a Myeloablative or Reduced-intensity Preparative Regimen Prior to HSCT for High-risk AML and MDS.
Description: Event-free survival at 6 months, where events are defined as relapse or death
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 15
Participants | 5 | 14

3. Primary Outcome: Number of Non-relapsed Deaths by 6 Months Post-transplant in Pediatric Patients Receiving a Myeloablative or Reduced-intensity Preparative Regimen Prior to HSCT for High-risk AML and MDS.
Description: Number of non-relapsed deaths that occur
Time Frame: Day 180
Population: Analysis population includes only subjects without relapse (i.e. subjects who relapse are therefore excluded from this analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 14
Participants | 1 | 0

4. Secondary Outcome: The Pace of Neutrophil Recovery
Description: Neutrophil Engraftment (the first of three consecutive days in which the absolute neutrophil count (ANC) exceeded 500/mcL)
Time Frame: Day of transplant to end of study (Day 365)
Measure: Median (Full Range); unit: Days
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 15
Days | 13 [9 to 18] | 13 [9 to 24]

5. Secondary Outcome: The Pace of Platelet Recovery
Description: Platelet Engraftment (the first of three consecutive days in which the platelet count exceeded 20,000/mm3 without platelet transfusions for the preceding 7 days)
Time Frame: Day of transplant to end of study (Day 365)
Measure: Median (Full Range); unit: days
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 15
days | 38 [25 to 41] | 32 [18 to 50]

6. Secondary Outcome: Number of Participants Developing Acute Graft Versus Host Disease (aGVHD) by Grade
Description: Grade 0: no stage 1-4 of any organ. Grade I: stage 1-2 skin rash (stage 1: <25%, stage 2: 25-50% body surface area affected by maculopapular rash), no gut or liver involvement.
  Grade II: stage 3 skin rash (>50% body surface area affected), or stage 1 GI involvement (10-19.9 mL/kg/day volume of diarrhea), or stage 1 liver involvement (2-3 mg/dL total bilirubin level).
  Grade III: stage 0-3 skin rash with stage 2-4 GI involvement (stage 2: 20-30 mL/kg/day, stage 3: >30 mL/kg/day volume of diarrhea, stage 4: severe abdominal pain with or without ileus and/or grossly blood stool) or stage 2-3 liver involvement (stage 2: 3-6 mg/dL, stage 3: 6-15 mg/dL total bilirubin level).
  Grade IV: stage 4 skin rash (generalized erythroderma with bullous formation) or stage 4 liver involvement (>15 mg/dL total bilirubin level).
Time Frame: Day of transplant to end of study (Day 365)
Population: Subjects must survive at least until 100 days post-transplant for evaluation for acute graft-versus-host disease, i.e. subjects who die before 100 days post-transplant are not evaluable and therefore excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 5 | 15
Participants
  No aGVHD (Grade 0) | 3 | 7
  aGVHD Grade I | 2 | 3
  aGVHD Grade II | 0 | 5
  aGVHD Grade III | 0 | 0
  aGVHD Grade IV | 0 | 0

7. Secondary Outcome: Number of Participants Developing Chronic Graft Versus Host Disease (cGVHD) by Grade
Description: Limited cGVHD: localized skin involvement and/or hepatic dysfunction due to cGVHD.
  Extensive cGVHD: one or more of the following: generalized skin involvement; liver histology showing chronic aggressive hepatitis, bridging necrosis, or cirrhosis; involvement of eye, minor salivary glands or oral mucosa based on biopsy, or any other target organ.
  Mild cGVHD: 1 or 2 organs involved with no more than score 1 plus lung score 0. Moderate cGVHD: 3 or more organs involved with no more than score 1, or at least one organ (not lung) with score 2, or lung score 1.
  Severe cGVHD: at least one organ with score 3, or lung score 2 or 3.
Time Frame: Day of transplant to end of study (Day 365)
Population: Subjects must survive at least until 365 days post-transplant for evaluation for chronic graft-versus-host disease, i.e. subjects who die before 365 days post-transplant are not evaluable and therefore excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 5 | 13
Participants
  No cGVHD | 3 | 8
  Limited cGVHD | 1 | 4
  Extensive cGVHD | 1 | 1
  Mild cGVHD | 2 | 4
  Moderate cGVHD | 0 | 0
  Severe cGVHD | 0 | 1

8. Secondary Outcome: Disease-free Survival (DFS)
Description: The number of subjects who are alive without relapse/leukemia
Time Frame: Day 100 and 180 post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 15
Participants
  Day 100 | 5 | 14
  Day 180 | 5 | 14

9. Secondary Outcome: Treatment-related Mortality (TRM)
Description: The number of subjects deceased due to transplant-related (i.e. non-relapse) causes
Time Frame: Day 100 and 180 post-transplant
Population: Subjects who die due to transplant-related causes by 100 and 180 days post-transplant, thus subjects who relapse before that time are excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 14
Participants
  Day 100 | 1 | 0
  Day 180 | 1 | 0

10. Secondary Outcome: The Number of Subjects With Overall Survival (OS)
Description: The number of subjects who are alive
Time Frame: Day 100 and 180 post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 15
Participants
  Day 100 | 5 | 15
  Day 180 | 5 | 14

11. Secondary Outcome: Day 0 Campath (Alemtuzumab) Level
Description: Campath (Alemtuzumab) level measured on the day of transplant
Time Frame: Day 0
Population: Only 2 subjects in Reduced-Intensity Conditioning arm and no subjects in Myeloablative Conditioning arm had a Day 0 Campath (Alemtuzumab) level drawn.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 2 | 0
mcg/mL | 0.24 [0.16 to 0.32] |

12. Secondary Outcome: Pace of Immune Reconstitution
Description: Immune recovery as measured by lymphocyte subsets
Time Frame: Day 180
Population: One subject in each arm did not survive to Day 180
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 5 | 14
cells/mm3
  CD3 Count (Total T-cells) | 405 [212 to 900] | 405 [122 to 2569]
  CD4 Count (Helper T-cell) | 171 [128 to 270] | 199.5 [56 to 733]
  CD8 Count (Suppressor T-cells) | 222 [65 to 577] | 113 [39 to 2067]
  CD19 Count (Total B-cells) | 347 [101 to 1615] | 366.5 [0 to 2022]
  CD16/56 Count (Total NK cells) | 359 [147 to 726] | 218 [25 to 1288]

13. Secondary Outcome: Incidence of Primary Graft Failure.
Description: The failure to achieve an ANC ≥500/μL after 42 days, determined by three consecutive measurements on different days, and not caused by recurrent leukemia.
Time Frame: Post-transplant to 42 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 15
Participants | 0 | 0

14. Secondary Outcome: Incidence of Grades 4 and 5 Adverse Events
Description: Adverse events as assessed by CTCAE
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 6 | 15
Participants
  White blood dell decreased | 6 | 15
  Platelet count decreased | 6 | 15
  Lymphocyte count decreased | 6 | 15
  Neutrophil count decreased | 6 | 12
  Sepsis | 1 | 6
  Anemia | 1 | 1
  Hyperglycemia | 1 | 0
  Alkaline phosphatase elevated | 0 | 1
  GGT increased | 1 | 0
  Febrile neutropenia | 0 | 1
  Pneumonitis | 1 | 0
  Pneumothorax | 1 | 0
  Bronchopulmonary hemorrhage | 1 | 0
  Multi-organ failure | 1 | 0
  Cardiac arrest | 1 | 0
  Encephalitis infection | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 180
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/15
Serious Adverse Events (participants affected / at risk) | 6/6 | 15/15
Other Adverse Events (participants affected / at risk) | 0/6 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced-Intensity Conditioning (N=6) | Myeloablative Conditioning (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Sinusoidal obstruction syndromw (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (4) | 10 (11)
Viremia (Infections and infestations) | 1 (2) | 2 (3)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (3)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) — Pneumonia
Upper respiratory infection (Infections and infestations) | 1 (1) | 3 (5)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 6 (6) | 15 (15) — Leukopenia
Platelet count decreased (Investigations) | 6 (6) | 15 (15) — Thrombocytopenia
Lymphocyte count decreased (Investigations) | 6 (6) | 15 (15) — Lymphopenia
Neutrophil count decreased (Investigations) | 6 (6) | 12 (12) — Neutropenia
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Low hemoglobin level
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Elevated blood glucose level
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Encephalitis infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT02626715/Prot_SAP_000.pdf